CLINICAL TRIAL: NCT02293759
Title: Prospective Non-randomized Trial Comparing Holmium Laser Enucleation of the Prostate Versus Greenlight Laser Photoselective Vaporization of the Prostate in Treating Benign Prostate Hyperplasia in Patients With Bleeding Tendency
Brief Title: Trial of HoLEP vs. PVP in Treating BPH in Patients With Bleeding Tendency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Dr, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mans-2014-04
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH- LASER- PROSTATE- BLEEDING TENDENCY
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HoLEP (Active Comparator): Holmium laser enucleation of the prostate
  Interventions: Procedure: HoLEP
- Greenlight laser PVP (Active Comparator): Phtoselective vaporization of the prostate
  Interventions: Procedure: Greenlight laser PVP

INTERVENTIONS:
Procedure: HoLEP — Holmium laser enucleation of the prsotate
  Arms: HoLEP
Procedure: Greenlight laser PVP — Greenlight laser (532nm) Photoslective vaporization of the prostate
  Arms: Greenlight laser PVP

SUMMARY:
Patients presented for BPH surgery at our out patient clinic will be assessed for abnormal bleeding profile.

Patients with bleeding tendency will be offered either HoLEP or Greenlight laser PVP based on prostate size cut off point of 80ml Larger prostates will be treated with HoLEP Smaller prostates will be treated with greenlight PVP

DETAILED DESCRIPTION:
Elderly patients with bleeding tendency either secondary;

1. Strict antiplatelet intake
2. Strict anticoagulant intake
3. uncorrected natural bleeding tendency e.g; patients with liver cell failure are at higher risk of perioperative bleeding when subjected to prostate surgery.

Laser prostate surery was introduced to overcome this difficulty. However, till now there is no head to head comparision of different types of laser procedures in treating this subset of patients In the current study patients presented for BPH surgery in a tertiarry referral prostate unit will be assessed for bleeding tendency and will be treated either by Holmium laser enucleatiuon of the prostate or Greenlight laser vaporization of the prostate Single surgeon will perform all cases

ELIGIBILITY:
Inclusion Criteria:

* BPH patients candidate for transurethral prostate surgery after failure of medical treatment
* Perioperative uncorrected Blleding tendency

  1. patients with naturally induced uncorrectable bleeding tendency;

     1. platelet count less than 100000/mm3
     2. INR more than 1.5
  2. Patients on oral antiplatlet that deemed unsafe to stop prior to surgery as per intenist
  3. Patients on oral anticoagulant that deemed unsafe to stop prior to surgery as per intenist

Exclusion Criteria:

* Correctable bleeding tendency

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
perioperative blood loss | 48 hours

SECONDARY OUTCOMES:
readmission | 30 days
blood transfusion | 30 days
flow rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed m Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt